CLINICAL TRIAL: NCT03856346
Title: Intraocular Lens Power Calculation for Combined Phaco-vitrectomy Procedures: Calculation of a New Constant for Biometry IOL-formulas
Brief Title: Intraocular Lens Power Calculation for Combined Phaco-vitrectomy Procedures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Josef Guber, Consultant ophthalmic surgeon, Cantonal Hospital of St. Gallen
Other Study IDs: Phaco-vity-biometry study
Record Dates: First submitted 2019-02-05; First posted 2019-02-27 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Intraocular Lens Calculation; Combined Phaco-vitrectomy
Keywords: Vitrectomy; Phacoemulsification; Biometry; IOL calculation; Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Phaco-vitrectomy
  Interventions: Diagnostic Test: Biometry

INTERVENTIONS:
Diagnostic Test: Biometry — Biometry for phaco-vitrectomy procedures pre- and postoperatively

SUMMARY:
The aim of the study is to evaluate the degree of refractive error postoperatively in combined procedures and to calculate a new constant in order to improve current state of the art biometry calculations.

DETAILED DESCRIPTION:
The IOL power calculation in combined phaco-vitrectomy has been performed similar to that in cataract surgery alone. In patients who undergo combined phaco-vitrectomy, deviations in refractive outcomes may be observed because of possible errors in measurement of axial length, changes in the properties of the vitreous cavity after removal of the vitreous, or intraocular tamponade. Most of the previous studies have reported variable degrees of myopic shift after phaco-vitrectomy for diabetic retinopathy, epiretinal membrane, and macular hole. Furthermore, use of intraoperative gas may increase further the risk of anterior displacement of the intraocular lens which may induce a higher myopic shift. However, these publications did not provide any quantification of the spherical deviations nor calculate any specific constant in order to improve currents state of art biometry calculations.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo a combined procedure with phacoemulsification and pars plana vitrectomy

Exclusion Criteria:

* Sulcus fixation of the IOL, sulcus suture of the IOL, or intra-scleral IOL fixation because of intraoperative posterior capsule rupture
* corneal disease, such as keratoconus, that interfered with refractive results
* IOL implantation with a toric IOL or multifocal IOL
* History of previous vitrectomy or corneal transplantation
* Other coexisting ocular disease such as proliferative diabetic retinopathy, advanced age-related macular degeneration, uveitis, acute retinal necrosis, Coat's disease, proliferative vitreous retinopathy, or trauma
* Intraocular tamponade using silicon oil

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who undergo a combined procedure with phacoemulsification and pars plana vitrectomy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Refractive prediction error (measured by subjective refraction, in diopters) | 6 weeks postoperatively
  postoperative actual subjective refraction minus preoperative planned refraction in spherical equivalence (in diopters)
Absolute prediction error (measured by subjective refraction, in diopters) | 6 weeks postoperatively
  absolute value of the difference between postoperative actual refraction and preoperative planned refraction (in diopters)
Changes in Axial Length (measured by biometry, in milimeters) | 6 weeks postoperatively
  Change of axial length postoperatively (in milimeter)
Changes in corneal curvature (measured by corneal topography, in diopters) | 6 weeks postoperatively
  change in corneal curvature (in diopters)

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital of Sankt Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No